CLINICAL TRIAL: NCT06076954
Title: Development, Feasibility and Acceptability of an Internet-based Cognitive Behavioral (iCBT) Intervention for Adolescents With Anxiety Disorders
Brief Title: Development, Feasibility and Acceptability of an iCBT Intervention for Adolescents With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CM1
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planned therapist feedback iCBT (Experimental): Participants in the planned therapist feedback iCBT condition will receive the iCBT intervention with planned feedback after each completed module. The therapist may spend a max. of 15 minutes giving feedback per module.
  Interventions: Behavioral: CoolMinds
- On-demand therapist feedback iCBT (Experimental): Participants in the on-demand therapist feedback iCBT condition will receive the intervention with on-demand feedback that is participant-initiated. The therapist may spend a max. of 15 minutes giving feedback per module.
  Interventions: Behavioral: CoolMinds

INTERVENTIONS:
Behavioral: CoolMinds — CoolMinds consists of 11 adolescent sessions and 9 parent sessions to be completed simultaneously during a 14-week treatment period. The main components comprise psychoeducation, cognitive restructuring, exposure therapy, and relapse prevention. The parent program also comprises information on how to handle school absenteeism for parents and teachers or pedagogues. The intervention is mainly transdiagnostic within the anxiety disorders but also includes diagnosis specific modules and content allowing for more personalized treatment. The treatment is delivered via a telephone app but can also be accessed via computer.
  Other Names: Internet-based cognitive behavioral therapy; Technology-delivered cognitive behavioral therapy; iCBT

SUMMARY:
The aim of the feasibility study is twofold: 1) to test the feasibility of the study design, and 2) to test the preliminary efficacy and the acceptability of a new iCBT intervention when delivered with different levels of therapist support. The feasibility trial will provide important information on the initial participant responses, and on how to properly collect data in the subsequent RCT.

The feasibility trial is conducted as a randomized study with 16 participants consisting of two conditions: 1) guided iCBT, and 2) on-demand iCBT, both to be completed over a 14-week period. Participants in the guided iCBT condition will receive the new iCBT intervention with planned feedback after each completed module. Participants in the on-demand iCBT condition will receive the intervention with on-demand feedback that is participant-initiated. In both conditions, the therapist may spend a max. of 15 minutes giving feedback per module. As there is no evidence on what amount of therapist support is sufficient for adolescents, the allowed time spent giving feedback will not differ between the two conditions in the feasibility trial. Thus, data on engagement will be collected to inform how the two treatment conditions differ. The trial includes data points at pre-treatment (T1) and post-treatment (T2) where the same measures will be administered as are planned in the RCT.

Acceptability of the intervention will be investigated by conducting semi-structured interviews with the participants. The interview will include an evaluation of the intervention, client satisfaction and potential reasons for drop out.

The results from the feasibility trial will be used to inform the subsequent RCT and to revise the intervention, procedures, and conditions if needed.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 17 years of age
* Primary anxiety diagnosis
* Must have the ability to read and write Danish
* Must have Internet access
* Must have a parent able to participate in the treatment alongside the adolescent

Exclusion Criteria:

* Specific phobia of blood-injection-injury type
* An autism spectrum disorder
* Psychotic symptoms
* Bipolar disorder
* Current suicidal ideation or self-mutilating behavior
* Current alcohol or substance abuse
* Moderate to severe depression
* Current eating disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The Youth Online Diagnostic Assessment (YODA) | Pre-intervention, post-intervention (12 weeks after commencing treatment)
  An online diagnostic assessment tool that assesses DSM-5 anxiety disorders and specific phobias. Each present diagnosis is assigned a clinician-rated severity score ranging from 0 (minimal/absent) to 4 (pervasive). Typically subclinical disorders would receive a rating of 0 or 1, and clinical disorders a rating of 1 to 4.
Spence Children's Anxiety Scale (SCAS-C/P) | Pre-intervention, post-intervention (12 weeks after commencing treatment)
  A 44-item self-report questionnaire assessing anxiety symptoms of six different anxiety disorders in DSM-IV: generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive compulsive disorder and physical injury fears. Symptoms are rated on a 4-point frequency scale ranging from 0 (never) to 3 (always) (min. = 0; max. = 114). A higher score indicates increased symptom severity. The Danish version has demonstrated good psychometric properties

SECONDARY OUTCOMES:
Child Anxiety Life Interference Scale (CALIS) | Pre-intervention, post-intervention (12 weeks after commencing treatment)
  CALIS measures the impact of youth anxiety on various areas of life functioning such as school, extracurricular activities, family life and friendships. Impact is reported on a 5-point severity scale ranging from 0 (not at all) to 4 (a lot) (min. = 0; max = 56). A summed score of all items is used to indicate level of impact, where a higher score indicates greater impairment. CALIS has shown satisfactory internal consistency and moderate test-retest reliability.
The Patient Health Questionnaire (PHQ-9) | Pre-intervention, post-intervention (12 weeks after commencing treatment)
  A 9-item questionnaire used to measure youth depressive symptoms and suicidal ideation within the past 2 weeks. Symptoms are rated on a frequency scale ranging from 0 (not at all) to 3 (nearly everyday). The symptoms are evaluated independently by adolescents. A summed score of all 9 items is used to indicate symptom severity (min. = 0; max. = 27), where a higher score indicates greater severity and possible presence of a depressive disorder.

OTHER OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | Post-intervention (12 weeks after commencing treatment)
  An 8-item questionnaire used to measure general satisfaction with a received treatment. Satisfaction is reported using a 4-point scale ranging from 1 (lowest degree of satisfaction) to 4 (highest degree of satisfaction). A summed score of all items is used to indicate level of satisfaction (min = 8; max. = 32). The scale has shown high internal consistency and concurrent validity.
EuroQol-5 Dimension Youth (EQ-5D-5L) | Pre-intervention, post-intervention (12 weeks after commencing treatment)
  A 5-item self-report questionnaire assessing quality of life and self-rated health. The items cover five domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety and depression. Each domain is assigned a score from 1 (no health problems) to 3 (a lot of health problems) and based on these scores, a unique health state can be identified for each participant.
Negative Effects Questionnaire (NEQ) | Post-intervention (12 weeks after commencing treatment)
  A 20-item questionnaire used to monitor the occurrence of negative effects in psychological treatments. Participants are asked to report whether specific things have occurred or not during treatment, how negatively it affected them, and whether the negative affect is attributed to the received treatment or other circumstances. The items can be summed together in order to get a frequency measure of the number of negative effects the respondents have experienced, divided by treatment or other circumstances. NEQ shows acceptable psychometric properties.
Systems Usability Scale (SUS) | Post-intervention (12 weeks after commencing treatment)
  A 10-item questionnaire used to assess the subjective experience of usability of a computer system. Participants are asked to score 10 different statements about the computer system on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree). A higher summed score indicates greater comfortability with the computer system. A Danish version of the SUS has been validated in a mental health care setting.
Engagement with the program: Wordcount | Post-intervention (12 weeks after commencing treatment)
  Number of words in the in-program text modules and number of words in messages sent by both participant and therapist.
Engagement with the program: number of logins | Post-intervention (12 weeks after commencing treatment)
  Number of logins in the digital platform.
Engagement with the program: Time spent on feedback | Post-intervention (12 weeks after commencing treatment)
  Therapist time spent giving feedback reported in minutes.
Demography | Pre-intervention
  Sociodemographic measures include participants' age and gender, and parents' level of education, and primary caregiver in case of single parents.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mathiasen, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen NM, Skaarnes H, Mathiasen K, McLellan LF, Thastum M, Lomholt JJ. Internet-based cognitive behavioral therapy (ICBT) for adolescents with anxiety disorders delivered with different types of therapist support: a randomized feasibility trial. Cogn Behav Ther. 2025 Jul 3:1-24. doi: 10.1080/16506073.2025.2522995. Online ahead of print. PMID 40607688